CLINICAL TRIAL: NCT04519905
Title: Phase III Study of Concurrent Radiotherapy in Elderly Patients With Esophageal Squamous Cell Carcinoma (ESO-Shanghai 15)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huadong Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Gansu Cancer Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Fujian Cancer Hospital (Other Government); Taihe Hospital (Other); Wuxi No. 4 People's Hospital (Other); Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai15
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Survival
Keywords: esophageal squamous cell carcinoma; elderly patients; chemoradiotherapy; definitive radiotherapy; survival
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemoradiotherapy (Experimental): 50.4Gy/28Fx; Paclitaxel plus carboplatin
  Interventions: Drug: Paclitaxel plus carboplatin; Radiation: radiotherapy
- radiotherapy (Active Comparator): 61.2Gy/34Fx
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: Paclitaxel plus carboplatin — Paclitaxel （45mg/m2) plus carboplatin (AUC=2); five cycles; qw
  Arms: chemoradiotherapy
Radiation: radiotherapy — Different radiotherapy dose in different groups.

SUMMARY:
So far, there is no specific clinical guideline for elderly patients (>75 yr) with esophageal squamous cell carcinoma (ESCC). Patients with locally advanced ESCC were enrolled and randomly assigned to either definitive radiotherapy group (61.2Gy/34Fx） or the chemoradiotherapy group (50.4Gy/28Fx；Paclitaxel plus carboplatin). The primary end point was 3-year overall survival (OS). The second end points included life quality, radiation side effects and 3-yr cancer specific survival.

DETAILED DESCRIPTION:
Up to now, definitive radiotherapy was major treatment plan for elderly ESCC patients. However, whether elective elderly patients can obtain survival benefits through chemoradiotherapy is not clear. Thus we design the clinical trail to answer the question.

Three hundred and twenty elderly patients with ESCC would be recruited. There are two stratification factors including 80 years old and lymph node metastasis. The patients in the chemoradiotherapy group were treated with paclitaxel (45mg/m2) and carboplatin (AUC=2) one cycle per week for five cycles.The primary end point was 3-year overall survival (OS). The second end points included life quality, radiation side effects and 3-yr cancer specific survival. The life quality questionnaire included QlQ-C30 and OES-18.

ELIGIBILITY:
Inclusion Criteria:

* Indicates no limit on eligibility based on the sex of participants
* The 76 years old for the minimum age a potential participant must meet to be eligible for the clinical study.
* Esophageal squamous cell carcinoma confirmed by pathology
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* Local advanced esophageal squamous cell carcinoma (T2-4N0-1M0-1a, TxN1M0-1a, TxNxM1a, TxNxM1b (M1b only for supraclavicular lymph node metastasis) (AJCC 6th)
* Use of an effective contraceptive for adults to prevent pregnancy
* No severely abnormal hematopoietic, cardiac, pulmonary, renal, or hepatic function
* No immunodeficiency
* ECOG 0-1.
* Life expectancy of more than 3 months.

Exclusion Criteria:

* Total radiotherapy dose cannot reach 61.2Gy/34Fx
* Esophageal perforation, or hematemesis
* History of radiotherapy or chemotherapy for esophageal cancer
* History of surgery within 28 days before Day 1
* History of prior malignancies (other than skin basal cell carcinoma or cervical carcinoma in situ with a disease-free survival of at least 3 years)
* Participation in other interventional clinical trials within 30 days
* Pregnant or breast-feeding women or fertile patients
* Drug addiction,
* alcoholism or AIDS
* Uncontrolled seizures or psychiatric disorders

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
overall survival difference of definitive radiotherapy and chemoradiotherapy groups | 3-year
  The time between the start of the study treatment (Day 1) and death from any cause or last follow-up for patients alive at the end of the study.

SECONDARY OUTCOMES:
difference of quality of life between different groups | the period of treatment within 7 weeks and follow up time with an average of 3months
  Assess the quality of life through life quality questionnaire.
radiation side effects | acute side effects within 3 months, late side effects for 3 months later
  Record the radiation side effects including acute and late side effects.
cancer specific survival | 3-year
  The time between the start of the study treatment (Day 1) and death from tumor or last follow-up for patients alive at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, doctor, Study Chair — Fudan University; Xiangpeng Zheng, doctor, Principal Investigator — Huadong Hospital
Locations (3):
- China (3):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No